CLINICAL TRIAL: NCT02823990
Title: Phase II Trial of TG4010 Plus Nivolumab in Previously Treated Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: TG4010 and Nivolumab in Patients With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Megan Daly, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Transgene (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Megan Daly, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 885316; UCDCC#263 (Other: UC Davis); UCDCC#263 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2016-00960 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage I Non-Small Cell Lung Cancer; Stage II Non-Small Cell Lung Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TG4010; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment TG4010 + nivolumab (Experimental): Patients receive TG4010 SC once per week for courses 1-3 and every 2 weeks for courses thereafter and nivolumab IV over 30 minutes every 2 weeks. Courses repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: TG4010; Biological: Nivolumab

INTERVENTIONS:
Biological: TG4010 — Given SC
  Other Names: Modified Vaccinia Ankara Encoding Human MUC-1 Antigen and Interleukin-2 Suspension; MVA-MUC1-IL2; MVA-MUC1-IL2 Vaccine
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well TG4010 and nivolumab work in previously treated patients with non-small cell lung cancer. Vaccines that are made from a gene-modified virus, such as TG4010, may help the body build an effective immune response to kill tumor cells. Monoclonal antibodies, such as nivolumab, interfere with the ability of tumor cells to grow and spread. Giving TG4010 and nivolumab together may work better in previously treated patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To evaluate the efficacy of nivolumab plus TG4010 (modified vaccinia virus Ankara [MVA]-human mucin 1 [MUC1]-interleukin-2 [IL2] vaccine) in previously treated patients with stage IV non squamous non-small cell lung cancer (NSCLC) with respect to objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OBJECTIVES:

Define the safety and toxicity profile of nivolumab plus TG4010 by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.

Determine progression-free survival by RECIST 1.1.

Determine overall survival.

Determine the duration of response and the occurrence of responses over time.

Determine the rate and duration of stable disease.

Determine the disease control rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-squamous NSCLC; patients with adenocarcinoma must have had epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) mutational testing; those with an actionable mutations/rearrangements are excluded
* Stage IIIB or IV patients must have progressed after a platinum based chemotherapy; a maximum of 3 previous systemic regimens are allowed (one regimen can be a tyrosine kinase inhibitor); patients with stage I-IIIB NSCLC who have progressed within 6 months of a full dose platinum based regimen as adjuvant therapy or with radiotherapy are eligible; patients who received weekly low dose chemotherapy with radiation only are not eligible
* At least one measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) based on RECIST version 1.1
* Performance status (PS) 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Minimum life expectancy of 3 months
* Hemoglobin >= 10.0 g/dL
* White blood cells (WBC) >= 3.0 x 10^9/L
* Neutrophils >= 1.5 x 10^9/L
* Total lymphocyte count >= 0.5 x 10^9/L
* Platelet counts >= 100 x 10^9/L
* Serum alkaline phosphatase =< 3 x upper limit of normal (ULN) in absence of liver or bone metastases and =< 5 x ULN in patients with documented bone or liver metastases
* Total bilirubin =< 1.5 x ULN
* Serum transaminases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) =< 2.5 x ULN in the absence of liver metastases and =< 5 x ULN in case of liver metastases
* Glomerular Filtration Rate >= 60 mL/min (according to Modification of Diet in Renal Disease [MDRD] formula or Cockcroft & Gault formula)
* Serum albumin >= 30 g/L
* Effective contraception during the study period and for 5 months after the last study treatment administration (male and female patient)
* Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients having active central nervous system (CNS) metastases; patients adequately treated and neurologically returned to baseline (except for residual signs of symptoms related to the CNS treated) for at least 2 weeks prior to enrolment are allowed; in addition, patients must be either off corticosteroids or on a stable or decreasing dose of < 10 mg daily prednisone or equivalent
* Prior exposure to cancer immunotherapy including any immune checkpoint inhibitor and/or cancer vaccines
* Prior history of other malignancy except:

  * Basal cell carcinoma of skin
  * Cervical intra-epithelial neoplasia
  * Other cancer curatively treated with no evidence of disease for at least 2 years
* Patients under chronic treatment with systemic corticosteroids or other immunosuppressive drugs (e.g. cyclosporine) for a period of at least 4 weeks and whose treatment was not stopped 1 week prior to start of the study treatment (day 1 [D1] of cycle 1)
* Positive serology for human immunodeficiency virus (HIV) or hepatitis C virus (HCV); presence in the serum of the antigen hemoglobin (HBs)
* Patient with any underlying medical condition that the treating physician considers might be aggravated by treatment or which is not controlled (e.g. elevated troponin or creatinine, uncontrolled diabetes)
* Patients with major surgery or radiotherapy within 4 weeks prior to the start of the study treatment (i.e. D1 of cycle 1); however, prior surgery or radiation therapy aimed at local palliation or attempted local disease control (except in case of thoracic radiotherapy) is permitted but has to be completed one week before treatment start
* Pregnant or nursing (lactating) women, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 10 mIU/mL); pregnancy is ruled out by a beta hCG test completed if necessary with an ultrasound
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are:

  * Women whose sexual orientation precludes intercourse with a male partner
  * Women whose partners have been sterilized by vasectomy or other means
  * Using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices [IUDs]; periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable)
* Patient with an organ allograft
* Known allergy to eggs, gentamicin, or platinum containing compounds
* Hypersensitivity to the active substance or to any of the excipients
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatment (i.e. D1 of cycle 1)
* Patient unable or unwilling to comply with the protocol requirements
* Subject has active, known or suspected autoimmune disease, including systemic lupus erythematodes, Hashimoto thyroiditis, scleroderma, polyarteritis nodosa, or autoimmune hepatitis
* Subject has any peripheral neuropathy >= National Cancer Institute (NCI) CTCAE grade 2 at enrollment
* Subject has a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies; any lung disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity
* History of any of the following cardiovascular conditions within 12 months of enrollment: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association
* Left ventricular ejection fraction (LVEF) less than the lower limit of normal (LLN) as assessed by echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kelly, Principal Investigator — University of California, Davis
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment TG4010 + nivolumab: Patients enrolled to receive TG4010 SC once per week for courses 1-3 and every 2 weeks for courses thereafter and nivolumab IV over 30 minutes every 2 weeks. Courses repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  TG4010: Given SC Nivolumab: Given IV
Period: Overall Study
Arm/Group | Treatment TG4010 + nivolumab
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment TG4010 + Nivolumab
Number analyzed (Participants) | 13
Age, Customized [Median (Full Range); unit: years] | 69 [56 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: ORR Defined as the Proportion of Patients Whose Best Overall Response (BOR) is Either Complete Response (CR) or Partial Response (PR) According to RECIST 1.1
Description: Number of patients with a best overall response of CR or PR, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Number; unit: Proportion of evaluable participants
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 12
Proportion of evaluable participants | 0.083

2. Secondary Outcome: Disease Control Rate (DCR) Defined as the Proportion of Patients Whose Best Overal Response is Either CR, PR or SD, Assessed by RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI. Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since the treatment started. Disease control rate (DCR) defined as the proportion of patients whose best overall response (BOR) is either CR, PR or SD,
Time Frame: Up to 4 years
Measure: Number; unit: Proportion of evaluable participants
Groups:
- Treatment TG4010 + nivolumab: Patients receive TG4010 SC once per week for courses 1-3 and every 2 weeks for courses thereafter and nivolumab IV over 30 minutes every 2 weeks. Courses repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity. TG4010: Given SC. Nivolumab: Given IV
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 12
Proportion of evaluable participants | 0.25

3. Secondary Outcome: Duration of Response (DOR) Defined as Patients Whose Best Overall Response is CR or PR (Confirmed Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI; Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Duration of response (DOR) defined as patients whose best overall response is CR or PR (confirmed response)
Time Frame: Time from the first documented response (CR or PR) until the event defined as first documented disease progression, assessed for up to 4 years
Population: Overall number of particpants analyzed = 1 (One participant had a documented response of CR or PR)
Measure: Mean (Full Range); unit: years
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 1
years | 4 [4 to 4]

4. Secondary Outcome: Number of Participants With Adverse Events Reported Per CTCAE v4.0
Time Frame: From the first dose to 100 days after last treatment, approximately up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 13
Participants | 13

5. Secondary Outcome: Overall Survival (OS)
Time Frame: Time from enrollment until death from any cause, assessed for up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 13
days | 220 [171 to 341]

6. Secondary Outcome: Progression Free Survival (PFS) Defined by RECIST 1.1
Description: Progression free survival (PFS) defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from enrollment to the date of first documented radiographic tumor progression or death due to any cause, whichever occurs first, assessed for up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 12
days | 41 [39 to 124]

7. Secondary Outcome: Stable Disease (SD) Rate Defined as the Proportion of Patients Whose Best Overall Response (BOR) is SD, Assessed by RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI; Stable disease (SD) rate defined as the proportion of patients whose best overall response (BOR) is stable disease (SD),
Time Frame: Up to 4 years
Measure: Number; unit: Proportion of evaluable participants
Arm/Group | Treatment TG4010 + nivolumab
Number analyzed (Participants) | 12
Proportion of evaluable participants | 0.17

ADVERSE EVENTS:
Time Frame: From the first dose to 100 days after last treatment. Approximately up to 2 years. All-Cause Mortality was from enrollment until death from any cause, assessed for up to 4 years
Arm/Group | Treatment TG4010 + nivolumab
All-Cause Mortality (participants affected / at risk) | 10/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment TG4010 + nivolumab (N=13)
Myocarditis (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment TG4010 + nivolumab (N=13)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blurred vision (Eye disorders) | 1
Chills (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Edema limbs (General disorders) | 2
Eye disorders - Other, Macular Edema (Eye disorders) | 1
Fatigue (General disorders) | 8
Fever (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flu like symptoms (General disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Injection site reaction (General disorders) | 8
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myocarditis (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 1
Non-cardiac chest pain (Gastrointestinal disorders) | 2
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Parainfluenza (Respiratory, thoracic and mediastinal disorders) | 1
Other, Brown Lesions on chest & back (Skin and subcutaneous tissue disorders) | 1
Other, Lesions on chest (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT02823990/Prot_SAP_000.pdf